CLINICAL TRIAL: NCT03129776
Title: Hyperpolarized 13C MR Imaging of Lactate in Patients With Locally Advanced Cervical Cancer for Treatment With Definitive Chemoradiation Therapy
Brief Title: Hyperpolarized 13C MR Imaging of Lactate in Patients With Locally Advanced Cervical Cancer (LACC) Cervical Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Lack of participants
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Ontario Institute for Cancer Research (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 355-2016
Record Dates: First submitted 2017-04-17; First posted 2017-04-26 (Actual); Last update posted 2022-09-22 (Actual); Status verified 2022-09

CONDITIONS: Uterine Cervical Neoplasms
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Fluorodeoxyglucose F18

STUDY DESIGN:
Intervention Model Description: Up to ten participants with newly diagnosed FIGO stage IB-IVA cervical cancer that are to receive definitive radiation with or without concurrent cisplatin, are to be recruited for this prospective single institutional study. Participants will receive a hyperpolarized carbon 13 MR spectroscopy and PET scan in addition to the standard imaging that is required for staging. A tumour biopsy will be obtained at the time of the initial clinic visit.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Hyperpolarized Pyruvate (13C) Injection (Active Comparator): Participants will be injected with the study drug Hyperpolarized Pyruvate (13C) Injection at a dose of 0.43 ml/kg and will have their cervix imaged using MRI.
  Interventions: Drug: Hyperpolarized 13C-Pyruvate
- 18F-FDG (Active Comparator): Participants will be injected with the study drug 18F-FDG at a dose of 5 MBq/kg to a a maximum of 500 MBq (megabecquerel) and will have their cervix imaged using PET-CT imaging.
  Interventions: Drug: 18F-FDG

INTERVENTIONS:
Drug: Hyperpolarized 13C-Pyruvate — The new imaging method being tested is called Metabolic MRI, which provides pictures of the metabolism occurring within cancer cells. It also involves injection of a contrast agent, Hyperpolarized Pyruvate (13C) Injection, into the arm vein. The participants will be injected with the study drug at a dose of 0.43 ml/kg and then receive a MRI scan.
  Arms: Hyperpolarized Pyruvate (13C) Injection
Drug: 18F-FDG — 18F-FDG is a radiopharmaceutical used in medical imaging. The uptake of 18F-FDG by tissues is a marker for the tissue uptake of glucose, which is correlated with certain types of tissue metabolism, particularly in cancer cells. The participant will be injected with the study drug at a dose of 5 MBq/kg to a maximum of 500 MBq and then receive a PET scan.
  Arms: 18F-FDG

SUMMARY:
The purpose of this study is to image tumour lactate in study participants with locally advanced cervical cancer. Our hypothesis is that lactate content in cervical tumours, as measured by hyperpolarized 13C Magnetic Resonance (MR) imaging, will correlate with diffusion-weighted MRI and 18FDG-PET (fluorodeoxyglucose-positron emission tomography). Furthermore, lactate imaging will potentially provide additional and more specific information regarding the metabolic activity of cervical tumours, thereby identifying regions of radiation resistance and guiding radiation treatment and brachytherapy.

DETAILED DESCRIPTION:
Patients with locally advanced cervical cancer can be offered definitive treatment with radiation therapy with concurrent chemotherapy for curative treatment. Brachytherapy is an essential part of this treatment, used to deliver high central doses after external beam radiation. Three-dimensional image-guided brachytherapy (3DIGBT) is gradually becoming the standard of care in many centres across the world. The use of Magnetic Resonance Imaging (MRI) or Computerized Tomography (CT) for planning helps ensure adequate coverage of tumours, minimizing doses to organs at risk. However, standard imaging modalities used in 3DIGBT typically include T2 and T1 weighted MRI sequences or CT scans and visualizing of the disease can often be challenging. Furthermore, it can be difficult to differentiate between active cervical cancer and fibrosis, leading to treatment of larger volumes when there is uncertainty (Akila contouring study).

High tumour lactate concentration has been linked to poor clinical outcomes in patients with solid tumours, including cervical cancers treated with radiation therapy [1, 2]. Three-dimensional imaging of tumour lactate in patients with locally advanced cervical cancers may be useful in identifying regions of radiation resistance and guiding treatment with chemoradiation and brachytherapy. The objective of this study is to image patients with locally advanced cervical cancer using hyperpolarized 13C MR imaging to obtain a measure of lactate levels in cervical tumours. Lactate images and measurements will be correlated with diffusion-weighted MRI, 18FDG-PET imaging and bioluminescence microscopy (BLI).

Up to ten participants with cervical cancer that are to receive radical treatment with radiation and possible concurrent cisplatin will be recruited for this study from Sunnybrook Health Sciences Centre (Sunnybrook). A snap-frozen biopsy of the tumour will be taken at the first clinic visit. Prior to treatment, baseline diffusion weighted MRI images and 18FDG-PET scans will be obtained. Hyperpolarized 13C MR imaging will be performed through the injection of 13C pyruvate and measurements of tumour lactate levels. Lactate levels will be correlated with measurements from bioluminescence microscopy. The images from hyperpolarized 13C MR imaging will also be compared to diffusion-weighted MR and 18FDG-PET images.

The purpose of this study is to image tumour lactate in study participants with locally advanced cervical cancer. Our hypothesis is that lactate content in cervical tumours, as measured by hyperpolarized 13C Magnetic Resonance (MR) imaging, will correlate with diffusion-weighted MRI and 18FDG-PET. Furthermore, lactate imaging will potentially provide additional and more specific information regarding the metabolic activity of cervical tumours, thereby identifying regions of radiation resistance and guiding radiation treatment and brachytherapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed squamous cell carcinoma, adenocarcinoma or adenosquamous carcinoma of the cervix, International Federation of Gynecology and Obstetrics (FIGO) stage IB-IVA
* Planned treatment with radical radiotherapy with or without concurrent cisplatin chemotherapy.
* Age ≥ 18 years.

Exclusion Criteria:

* Any anticancer treatment for their cervical cancer.
* Eastern Cooperative Oncology Group (ECOG) performance status > 2
* Other cervical cancer tumor histologies (e.g. small cell, serous)
* Contraindications to 18FDG PET-CT
* Inability to lie supine for 18FDG PET-CT
* Contraindication to radiotherapy (e.g. severe Crohn's disease)
* History of another invasive malignancy, except for non-melanoma skin cancer or tumors curatively treated with no evidence of disease for ≥ 5 years.
* Known pregnancy or lactating

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only biological females with a cervix will be recruited.
Enrollment: 4 (Actual)
Dates: Start 2017-11-13 (Actual); Primary Completion 2022-09-15 (Actual); Study Completion 2022-09-15 (Actual)

PRIMARY OUTCOMES:
Time resolved, 3D 13C lactate images from subjects with cervical cancer. | 1 year
  Feasibility of acquiring time resolved, 3D 13C lactate images from subjects with cervical cancer.

SECONDARY OUTCOMES:
Correlation of MRI and 18FDG-PET images | 1 Year
  Visual analysis and correlation between images obtained following Hyperpolarized Pyruvate (13C) Injection and 18FDG-PET imaging to identify cervical cancer.

CONTACTS AND LOCATIONS:
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No